CLINICAL TRIAL: NCT05520541
Title: Investigation of the Effects of Clinical Based LSVT-BIG Training and Home Based LSVT-BIG Training on Balance and Gait in Parkinson's Patients
Brief Title: The Effectiveness of LSVT-BIG Training in Improving Balance and Gait in Parkinson's Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sefa Eldemir, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3- PD-LSWT-Trainig
Record Dates: First submitted 2022-08-24; First posted 2022-08-30 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; LSVT-BIG Training; Home Based Exercise; Balance; Walking
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Two groups as clinical group and home group
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Group (Experimental): This group will receive clinical-based LSVT-BIG training
  Interventions: Other: Exercise
- Home Group (Active Comparator): This group will receive home-based LSVT-BIG training
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Both groups will receive exercise-based training

SUMMARY:
Parkinson's disease (PD) is a chronic, progressive disease that causes motor and non-motor symptoms due to dopaminergic neuron loss. Today, the treatment of PD in addition to optimal medical and surgical treatments, physiotherapy and rehabilitation approaches have an important place in the treatment. Recently, it has been stated that intensive rehabilitation interventions in the field of physiotherapy and rehabilitation can be more effective than traditional rehabilitation approaches. Lee Silverman VoiceTreatment- BIG (LSVT-BIG) is a high-intensity exercise model aimed at improving bradykinesia and hypokinesia in PD. There are many studies showing improvements in balance, walking, motor performance, reaching ability, postural control, quality of life and cognitive status after LSVT-BIG training in PD. However, it is seen that there is no study investigating the effect of LSVT-BIG training directly by applying it as a home program. For this reason, there is a need for studies investigating whether this intensive treatment method can be an alternative to the clinical environment by applying it as a home program.

DETAILED DESCRIPTION:
This study is planned as a randomized control trial. Patients will be randomly divided into two groups a clinical group and a home group. The clinical group will be received LSVT-BIG training four times a week for four weeks in the clinic. The home group will be received LSVT-BIG training two times a week for four weeks at the home and two times a week for four weeks at the clinical.

All assessments will be done before and after the 4-week intervention program or waiting period. The demographic characteristics of the participants initially will be taken. The outcome measures are balance and gait assessments.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age
* Having diagnosed with "Parkinson's Disease" by a specialist physician
* Having between 1-3 stages according to the Hoehn and Yahr Scale
* Mini-Mental Test score more than or equal 24

Exclusion Criteria:

- Any orthopedic, vision, hearing, cardiovascular, or perception problems that may affect the research results

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-07-22 (Actual)

PRIMARY OUTCOMES:
Static Balance- Baseline | Assessment will be conducted before the intervention.
  Assessment will be made with the Biodex Balance System
Static Balance- Post intervention | Assessment will be conducted immediately after the intervention.
  Assessment will be made with the Biodex Balance System
Gait speed- Baseline | Assessment will be conducted before the intervention.
  Assessment will be made with the BTS G-WALK, (BTS SpA, Via della Croce Rossa, 11 Padova, Italy;SN: 0213- 0378) during gait
Gait speed- Post intervention | Assessment will be conducted immediately after the intervention.
  Assessment will be made with the BTS G-WALK, (BTS SpA, Via della Croce Rossa, 11 Padova, Italy;SN: 0213- 0378) during gait
Gait cadence- Baseline | Assessment will be conducted before the intervention.
  Assessment will be made with the BTS G-WALK, (BTS SpA, Via della Croce Rossa, 11 Padova, Italy;SN: 0213- 0378) during gait
Gait cadence- Post intervention | Assessment will be conducted immediately after the intervention.
  Assessment will be made with the BTS G-WALK, (BTS SpA, Via della Croce Rossa, 11 Padova, Italy;SN: 0213- 0378) during gait

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Güçlü-Gündüz, PT, PhD., Study Director — Professor
Locations (1):
- Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to make PD data but when the statistical analysis of all data is made, all results will be shared.

REFERENCES:
- [Result] Millage B, Vesey E, Finkelstein M, Anheluk M. Effect on Gait Speed, Balance, Motor Symptom Rating, and Quality of Life in Those with Stage I Parkinson's Disease Utilizing LSVT BIG(R). Rehabil Res Pract. 2017;2017:9871070. doi: 10.1155/2017/9871070. Epub 2017 Feb 26. PMID 28331638
- [Result] Hirakawa Y, Takeda K, Koyama S, Naoi Y, Matsushita T, Nagai T, Motoya I, Sakurai H, Kanada Y, Kawamura N, Kawamura M, Tanabe S. Effect of Lee Silverman Voice Treatment (LSVT)(R) BIG on motor symptoms in a patient with severe Parkinson's disease: a case report. Physiother Theory Pract. 2022 Nov;38(13):3159-3168. doi: 10.1080/09593985.2021.1938304. Epub 2021 Jun 14. PMID 34125001